CLINICAL TRIAL: NCT01707095
Title: Bundling and Unbundling the Laparoscopic Electrosurgery Cord With the Camera Cord: A Randomized, Controlled Trial
Brief Title: Bundling and Unbundling the Laparoscopic Electrosurgery Cord With the Camera Cord
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 12-0906
Record Dates: First submitted 2012-09-21; First posted 2012-10-15 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Fatigue
Keywords: Electrosurgery; Radiofrequency energy; Monopolar instruments; Capacitive coupling; Thermal injury; Surgical complications
MeSH Terms: conditions — Fatigue; Hyperthermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bundling of cords (Experimental): The cords from the camera/active electrode will be bundled together along their lengths during a laparoscopic cholecystectomy.
  Interventions: Other: Bundling of cords
- Unbundling of cords (Experimental): The active electrode and camera cords will be place off opposite sides of the table and will not run adjacent to or in parallel with one another
  Interventions: Other: Unbundling of cords

INTERVENTIONS:
Other: Unbundling of cords — The active electrode and camera cords will be place off opposite sides of the table and will not run adjacent to or in parallel with one another
  Arms: Unbundling of cords
Other: Bundling of cords — The cords from the camera/active electrode will be bundled together along their lengths during a laparoscopic cholecystectomy.
  Arms: Bundling of cords

SUMMARY:
Electrosurgery is used in virtually every laparoscopic operation performed. Capacitive coupling is a common electrosurgery complication. Previous work biopsying the skin adjacent to laparoscopic port sites is a method to determine if capacitive coupling thermal injury to the skin occurs during a laparoscopic operation. [Willson et al. Surg Endosc (1997) 11:653] In our previous study, COMIRB 09-0049, we found thermal injury at 55% of umbilical trocar site skin biopsies and 35% of epigastric trocar site skin biopsies following laparoscopic cholecystectomy. Our benchtop research compared bundling of the camera cord with the active electrode cord versus unbundling of the camera cord with the active electrode cord and found a 59% decrease in heat generated in the unbundling experimental set-up. [Jones, EL, Robinson, TN, et al. Surg Endosc (2012) Epub.]

This study plans to compare thermal injury which occurs during two commonly used operating room set-ups. First, laparoscopic cholecystectomy with bundled camera/active electrode cords. And second, laparoscopic cholecystectomy with unbundled camera/active electrode cords. The primary outcome is the incidence of thermal injury at the skin adjacent to the camera port site (the umbilical port) that will be diagnosed by histology.

DETAILED DESCRIPTION:
We hypothesize that the unbundling of camera and active electrode cords will reduce the incidence of capacitive coupling thermal injuries to the skin adjacent to the camera port site in comparison to bundled active electrodes/camera cords during laparoscopic cholecystectomy operations.

SPECIFIC AIMS:

1. Compare incidence of skin burns by histology at the camera port site (umbilical port site) with bundled active electrode/camera cords to unbundled active electrode/camera cords.
2. Compare incidence of skin burns by histology at the active electrode port site (epigastric port site) with bundled active electrode/camera cords to unbundled active electrode/camera cords.
3. Compare incidence of skin burns by histology at the assistant port site with bundled active electrode/camera cords to unbundled active electrode/camera cords.

OUTCOME MEASURE:

Histologic evidence of thermal injury at the skin biopsy sites of the active electrode port, the camera port and the medial assistant port.

POPULATION TO BE ENROLLED:

Subjects undergoing elective cholecystectomy will be recruited in pre-operative clinic. All subjects will be 18 years and older.

STUDY DESIGN AND METHODS:

Written informed consent will be obtained in all subjects prior to enrollment. Subjects will be randomized on the day of surgery to undergo the laparoscopic cholecystectomy operation with either the bundled or unbundled camera and active electrode cords. The randomization process will occur by a random number generator. A total of 84 subjects will be recruited; 42 subjects per group. Shave skin biopsies will be performed at the lower edge of the incisions of the active electrode port, the camera port and the medial assistant port. The incisions and skin will be otherwise opened and closed in the routine clinical manner. The biopsy specimens will be analyzed for thermal injury by a blinded pathologist.

The incidence of skin burns created bundled or unbundled camera and active electrode cords will be compared individually at all three port sites by a blinded pathologist for histologic evidence of thermal injury.

Statistical analysis using a chi-squared test will be comparing the incidence of thermal injury at the each biopsy site for subjects with and without bundled cords. The primary outcome variable is thermal injury of skin at the umbilical trocar site, which is the camera trocar.

Baseline demographic information will be recorded on all patients: age, gender, BMI, operating room time, pre-op diagnosis, gallbladder histology, blood loss, and need to convert to open surgery.

SAMPLE SIZE CALCULATION:

The incidence of skin burns at the umbilical trocar site with bundled cords was 55% (11/20) in our previous study. Our prior benchtop research found that bundled cords resulted in an increase of temperature of 38.2°C at the tip of the telescope in comparison to a 15.7°C increase in temperature with separated cords. This finding suggests that 41% (15.7/38.2) of the heat is produced when the camera cord is unbundled from the active electrode cord in comparison to when the cords are bundled. This data is used to estimate that the unbundled cord group will have an incidence of thermal injury of 23% (0.41 x 55%).

Power 80% A sample size calculation comparing proportions was performed which compared 0.55 (bundled cords) incidence of thermal injury versus 0.23 (unbundled cords) incidence of thermal injury. A sample size of 36 per group has the power (1-β) 0.80 to detect a difference assuming α=0.05. We estimate a 15% dropout rate (this would be individuals who between their consent in pre-operative clinic and their operation decide to withdraw from the study). A 15% dropout rate is conservative in light of our prior experience recruiting similar patients when 0% (0/40) of individuals dropped out. Total sample size is estimated to be 72 (36 for each of two groups) plus 11 (15% dropout) for a total of 84 subjects.

STATISTICAL ANALYSIS:

The incidence of thermal injury to the skin (dichotomous variable) in the groups that had unbundled or bundled camera/active electrode cords will be compared using the Fischer's exact chi squared test.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older planned to undergo an elective laparoscopic cholecystectomy.

Exclusion Criteria:

* Patients undergoing urgent or emergent laparoscopic cholecystectomy operations
* Patients younger than 18

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas N Robinson, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

REFERENCES:
- [Background] Willson PD, van der Walt JD, Moxon D, Rogers J. Port site electrosurgical (diathermy) burns during surgical laparoscopy. Surg Endosc. 1997 Jun;11(6):653-4. doi: 10.1007/s004649900414. PMID 9171127
- [Background] Wu MP, Ou CS, Chen SL, Yen EY, Rowbotham R. Complications and recommended practices for electrosurgery in laparoscopy. Am J Surg. 2000 Jan;179(1):67-73. doi: 10.1016/s0002-9610(99)00267-6. PMID 10737583
- [Background] Jones EL, Robinson TN, McHenry JR, Dunn CL, Montero PN, Govekar HR, Stiegmann GV. Radiofrequency energy antenna coupling to common laparoscopic instruments: practical implications. Surg Endosc. 2012 Nov;26(11):3053-7. doi: 10.1007/s00464-012-2312-6. Epub 2012 May 12. PMID 22580879
- [Derived] Robinson TN, Jones EL, Dunn CL, Dunne B, Johnson E, Townsend NT, Paniccia A, Stiegmann GV. Separating the Laparoscopic Camera Cord From the Monopolar "Bovie" Cord Reduces Unintended Thermal Injury From Antenna Coupling: A Randomized Controlled Trial. Ann Surg. 2015 Jun;261(6):1056-60. doi: 10.1097/SLA.0000000000000841. PMID 26291952

RESULTS

PARTICIPANT FLOW:
Groups:
- Bundled: Active electrode cord and camera cord parallel
- Unbundled / Separated: Active electrode cord and camera cord separated
Period: Overall Study
Arm/Group | Bundled | Unbundled / Separated
Started | 42 | 42
Completed | 42 | 42
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bundling of Cords | Unbundling of Cords | Total
Number analyzed (Participants) | 42 | 42 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (15) | 44 (18) | 44 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 32 | 69
  Male | 5 | 10 | 15
Region of Enrollment [Number; unit: participants]
  United States | 42 | 42 | 84

OUTCOME MEASURES:

1. Primary Outcome: Histologic Thermal Injury to Umbilical Port Site Skin
Description: Shave biopsy of skin at the umbilical port site after elective laparoscopic cholecystectomy will be performed. The primary outcome is histologic evidence of burn at these port sites.
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Bundled | Unbundled / Separated
Number analyzed (Participants) | 42 | 42
participants | 24 | 13

2. Secondary Outcome: Histologic Evidence of Burn at the Epigastric Port Site Skin.
Description: Shave biopsy of skin at the epigastric port site after elective laparoscopic cholecystectomy will be performed. The secondary outcome is histologic evidence of burn at this port site.
Time Frame: 1 day
Measure: Number; unit: participants
Arm/Group | Bundled | Unbundled / Separated
Number analyzed (Participants) | 42 | 42
participants | 8 | 11

ADVERSE EVENTS:
Arm/Group | Bundled | Unbundled / Separated
Serious Adverse Events (participants affected / at risk) | 0/42 | 0/42
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bundled (N=42) | Unbundled / Separated (N=42)
(Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No